CLINICAL TRIAL: NCT07108816
Title: A Single-center, Phase II Clinical Trial Evaluating the Efficacy of Sacituzumab Tirumotecan in Combination With Tagitanlimab as Neoadjuvant Therapy for PD-L1-positive, Resectable Stage II to IIIB Non-small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-277
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Resectable Stage II-IIIB NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perioperative immunotherapy group (Experimental): Neoadjuvant Sacituzumab tirumotecan + tagitanlimab Followed by adjuvant tagitanlimab
  Interventions: Drug: Neoadjuvant Sacituzumab tirumotecan + tagitanlimab Followed by adjuvant tagitanlimab

INTERVENTIONS:
Drug: Neoadjuvant Sacituzumab tirumotecan + tagitanlimab Followed by adjuvant tagitanlimab — Patients will receive 4 cycles of neoadjuvant treatment with preoperative Sacituzumab tirumotecan in combination with tagitanlimab, followed by surgery.
  After surgery, patients will receive up to 13 cycles of adjuvant tagitanlimab.

SUMMARY:
In recent years, substantial progress has been made in the development of perioperative immunotherapy for non-small cell lung cancer (NSCLC). Accumulating evidence indicates that both neoadjuvant and adjuvant immunotherapy can significantly enhance key clinical endpoints, including pathological response rate, event-free survival (EFS), and disease-free survival (DFS), particularly in patients with stage II-III NSCLC. However, in the subset of patients with resectable stage II-IIIB NSCLC, the pathological complete response (pCR) rate following neoadjuvant immunotherapy remains modest at approximately 17-25%, underscoring the need for more effective therapeutic strategies and novel combination regimens. TROP2-targeted antibody-drug conjugates (TROP2-ADCs) have demonstrated promising antitumor activity and a manageable safety profile in patients with previously treated advanced NSCLC. Furthermore, the combination of Sacituzumab tirumotecan and tagitanlimab has shown robust efficacy in the first-line treatment of PD-L1-positive (tumor proportion score [TPS] ≥ 1%), driver gene-negative advanced NSCLC, with an objective response rate (ORR) exceeding 80%. Based on these encouraging data, we designed this study to evaluate the efficacy and safety of Sacituzumab tirumotecan in combination with tagitanlimab as neoadjuvant therapy in patients with PD-L1-positive (TPS ≥ 1%), resectable stage II-IIIB NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of informed consent signing.
2. ECOG performance status score of 0 or 1 within 7 days before administration.
3. Non-small cell lung cancer (NSCLC) confirmed by histological or cytological analysis.
4. Negative for EGFR sensitive mutations (no exon 19 deletion or exon 21 L858R substitution mutation) and negative for ALK fusion gene;
5. Positive PD-L1 expression (tumor proportion score [TPS] ≥ 1%) confirmed by immunohistochemistry (IHC).
6. No prior local treatment (e.g., surgery or radiotherapy) for non-small cell lung cancer (NSCLC) and no history of systemic anti-tumor therapy, including cytotoxic therapy, targeted therapy (such as tyrosine kinase inhibitors or monoclonal antibodies), cell therapy, immunotherapy, traditional Chinese medicine-based treatments, or any other investigational drug therapies.
7. Patients with resectable stage II-IIIB NSCLC (according to the 8th edition of the UICC/AJCC TNM staging system) after MDT evaluation;
8. At least one measurable lesion present, as defined by RECIST 1.1 criteria.
9. Patients willing to receive curative-intent surgical treatment.
10. Assessment by a surgeon confirms tumor resectability and absence of surgical contraindications.
11. Adequate organ and bone marrow function(with no receipt of blood transfusions, recombinant human thrombopoietin, or colony-stimulating factors within two weeks prior to first drug administration), defined as follows:

    1. Blood routine: Neutrophil count (NEUT#) ≥ 1.5×109/L; Platelet (PLT) ≥100×109/L; Hemoglobin ≥ 90g/L.
    2. Liver function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 times the upper limit of normal (ULN); total bilirubin (TBIL) ≤ 1.5 times ULN;
    3. Renal function: Ccr ≥ 60 ml/min (Cockcroft-Gault formula provided).
    4. International Normalized Ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) values are ≤ 1.5 times the upper limit of normal (ULN).
    5. Cardiac function: LVEF ≥ 50% by ECHO or MUGA scan.
12. For female subjects of childbearing potential and male subjects with reproductive potential, a commitment to effective medical contraception is required from the date of informed consent signing through 6 months after the last dose administration.
13. The subjects voluntarily joined this study, signed the informed consent form, and were able to comply with the visit and related procedures as stipulated in the protocol.

Exclusion Criteria:

1. Histological or cytological confirmation demonstrating the presence of small cell lung cancer, neuroendocrine carcinoma, or carcinosarcoma components within the tumor.
2. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies, or any other agent specifically targeting T-cell co-stimulatory or checkpoint pathways.
3. Prior treatment with TROP2-targeted therapy and/or topoisomerase I inhibitors.
4. Subjects requiring the use of strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) within 2 weeks prior to first dosing and throughout the study period are excluded (the use of strong CYP3A4 inhibitors or inducers is prohibited in this study; a list of representative CYP3A4 inhibitors and inducers can be found in Appendix 6). All subjects must avoid concomitant administration of any known drugs, herbal supplements, and/or dietary items that may induce CYP3A4 activity.
5. A history of other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin.
6. Known history of allergy to the study drugs or their components, immunodeficiency, or organ transplantation;
7. A history of interstitial lung disease (ILD) or non-infectious pneumonia requiring corticosteroid therapy, or current ILD or non-infectious pneumonia, or suspected ILD or non-infectious pneumonia at screening that cannot be ruled out by imaging; clinically significant pulmonary impairment due to concurrent lung conditions, including but not limited to underlying pulmonary disorders (e.g., pulmonary embolism within 3 months prior to study entry, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion), autoimmune, connective tissue, or inflammatory disorders with potential pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis), or prior pneumonectomy.
8. Active autoimmune diseases requiring systemic therapy within the past two years (hormone replacement therapy is excluded from systemic treatment, including conditions such as type 1 diabetes, hypothyroidism managed with thyroid hormone replacement alone, and adrenal or pituitary insufficiency treated solely with physiological doses of glucocorticoid replacement therapy).
9. Active infections requiring systemic treatment within 2 weeks prior to the first dose administration;
10. Active hepatitis B [positive hepatitis B surface antigen (HBsAg), with HBV-DNA testing required; HBV-DNA ≥ 500 IU/mL or above the lower limit of quantification (whichever is higher)] or hepatitis C (positive hepatitis C antibody and HCV-RNA above the lower limit of detection). Note: Subjects who are HBsAg-positive must receive anti-hepatitis B virus therapy during the study treatment period.
11. Positive serology for human immunodeficiency virus (HIV) or a history of acquired immune deficiency syndrome (AIDS); known active syphilis infection;
12. Concomitant diseases that, in the investigator's judgment, pose a significant risk to patient safety or may interfere with study completion, including but not limited to medication-uncontrolled hypertension, severe diabetes, or active infections.
13. A documented history of severe dry eye syndrome, severe meibomian gland dysfunction and/or blepharitis, or corneal disorders associated with delayed corneal healing;
14. Pregnant or breastfeeding women;
15. Any condition that may interfere with the assessment of the investigational drug, compromise subject safety, or affect the interpretation of study results, as well as any other condition that the investigator considers unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | Assessment of postoperative pathology within 6 weeks of neoadjuvant therapy
  0% residual viable tumor cells in the primary tumor and sampled lymph nodes

SECONDARY OUTCOMES:
Major Pathological Response | Assessment of postoperative pathology within 6 weeks of neoadjuvant therapy
  Major Pathological Response (≤10% residual viable tumor cells in the primary tumor and sampled lymph nodes)
R0 Resection Rate | Pre-operation
  The pathological results will showed that the incision margin was negative and no residual cancer cells were found under the microscope.
Objective Response Rate (ORR) | 1 month after surgery
  Defined as the proportion of patients whose tumor size shrinks to predefined values，which including cases of CR and PR. Objective tumor response will be assessed using RECIST 1.1. Subjects must have measurable tumor lesions at baseline, and the response evaluation criteria are classified as complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to RECIST 1.1.
Event-free survival(EFS) | Up to 24 months
  Defined as the time from treatment initiation to the first occurrence of any of the following events: disease progression precluding surgical treatment, local or distant recurrence, or death from any cause, assessed according to RECIST v1.1.
Overall survival (OS) | Up to 5 years
  Defined as the time from the initiation of study protocol treatment to the subject's death from any cause.
Adverse Events (AEs) | From date of treatment allocation until surgery or within 30 days after last dose of preoperative treatment
  The number of participants experiencing an AE will be assessed